CLINICAL TRIAL: NCT03527901
Title: Evaluation of Active Matrix Metalloproteinase-8 (aMMP-8) Chair-side Test in Different Periodontal Disease and Healthy Implants
Brief Title: Active Matrix Metalloproteinase-8 (aMMP-8) Chair-side Test in Different Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Veli Özgen Öztürk, Principal Investigator, Aydin Adnan Menderes University
Other Study IDs: BAP-17/1
Record Dates: First submitted 2018-05-05; First posted 2018-05-17 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2016-05

CONDITIONS: Periodontal Diseases
Keywords: aggressive periodontitis; healthy peri-implant; chairside test; chronic periodontitis
MeSH Terms: conditions — Periodontal Diseases; Aggressive Periodontitis; Chronic Periodontitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Chronic periodontitis: This groups participant has radiographically moderate alveolar bone loss, CAL > 5 mm and PD >6 mm in several sites of each quadrant
  Interventions: Diagnostic Test: GCF collection with aMMP-8 chair side test; Other: Saliva collection
- Generalized aggressive periodontitis: This demonstrated a generalized pattern of severe breakdown and CAL > 5 mm and PD > 6 mm on 8 > teeth; minimum three of those were other than first incisors or first molars
  Interventions: Diagnostic Test: GCF collection with aMMP-8 chair side test; Other: Saliva collection
- Gingivitis: This group has varying degrees of gingival inflammation, with CAL < 2 mm, without any radiographical bone loss due to periodontitis
  Interventions: Diagnostic Test: GCF collection with aMMP-8 chair side test; Other: Saliva collection
- Implant: Implants classified PD < 5 mm, no bleeding on probing, no suppuration and no radiographic bone loss > 0.5 mm
  Interventions: Diagnostic Test: GCF collection with aMMP-8 chair side test; Other: Saliva collection
- Health: Probing depth (PD) < 3mm, no gingival recession due to periodontal disease, and clinical attachment level (CAL) < 2 mm, BOP in < 10% of full-mouth score examination
  Interventions: Diagnostic Test: GCF collection with aMMP-8 chair side test; Other: Saliva collection

INTERVENTIONS:
Diagnostic Test: GCF collection with aMMP-8 chair side test
Other: Saliva collection

SUMMARY:
The aim of this study to evaluate the diagnostic accuracy of a new qualitative aMMP-8 POC test in different periodontal health and disease and as compared to the established quantitative laboratory method (ELISA)

DETAILED DESCRIPTION:
MMP-8 has been reported to reflect the inflammatory status in periodontal tissues and, therefore represent as potential biomarkers of periodontitis. A positive aMMP-8 test could be an early indicator of these excessive and undesired tissue reactions.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Nonsmokers

Exclusion Criteria:

* Participants were not included if they had systemic disease such as diabetes, cardiovascular.
* Participants who took regular medications that could affect of periodontal tissue
* Participants who received antibiotics less than 10 weeks before the study

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: All participants have minimum 20 teeth
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
aMMP-8 levels of GCF | 2 hours
  GCF levels measured by IFMA

SECONDARY OUTCOMES:
Salivary MMP-8 levels | 2 hours
  Saliva levels measured by IFMA